CLINICAL TRIAL: NCT00657488
Title: Multicenter, Randomized Study Comparing the Efficacy and Safety of Two Doses of Thalidomide (100 mg/Day Versus 400 mg/Day) in the Treatment of Subjects With Refractory or Relapsed Multiple Myeloma.
Brief Title: Thalidomide 100 mg/Day Versus Thalidomide 400 mg/Day in Relapse Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LATH0102/IFM0102
Record Dates: First submitted 2008-04-07; First posted 2008-04-14 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma, Thalidomide, dose, dexamethasone
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Thalidomide 100mg/day. Dexamethasone is administered at a dose of 40 mg/d, on 4 consecutive days (D1 - D4), with one course every four week in case of stable disease after 12 weeks of treatment or in case of Disease Progression
  Interventions: Drug: Thalidomide
- B (Active Comparator): Thalidomide 400mg/day. Dexamethasone is administered at a dose of 40 mg/d, on 4 consecutive days (D1 - D4), with one course every four week in case of stable disease after 12 weeks of treatment or in case of Disease Progression
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 100mg/day or 400 mg/day at bed time during one year
  Other Names: THALOMID

SUMMARY:
The objective of this study is to show that thalidomide at a dose of 100 mg/d (with remedial treatment with dexamethasone if a progression occurs) is equivalent in terms of efficacy with thalidomide at 400 mg/d (with remedial treatment with dexamethasone if a progression occurs) in the treatment of refractory or relapsed multiple myeloma after at least two courses of treatment. The use of thalidomide at 100 mg/d should reduce the side effects and improve the safety of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years who has been informed about the potential risks and side effects of the treatment and having signed an informed consent to take part in the various aspects of the study.
* Having a refractory or relapsed multiple myeloma after at least two courses of treatment.
* The patients with a refractory or relapsed multiple myeloma after a single course of treatment that included an alkylating drug, can be included if there is no alternative treatment.
* Concerning the thalidomide: Agreement to use and introduction of effective contraception by all the patients:

  1. For women of childbearing potential

     * Oral estroprogestogen contraception introduced at least 1 month before the first administration of thalidomide, and continued until the first menstruation following the end of the treatment, and their partners use a condom.
     * Qualitative serum test for beta-HCG negative: to be done on Day 2 or 3 of the menstrual cycle just before the 1st prescription of thalidomide; in a context of spaniomenorrhea or amenorrhea the test should be done within 3 days after the 1st prescription of thalidomide.
  2. For post-menopausal women

     * 1st situation: Known sterility due to:

       * total hysterectomy;
       * total ovariectomy;
       * total salpingectomy
     * 2nd situation: Natural menopause

       * amenorrhea for at least 1 year and
       * negative progestagen test and
       * plasma FSH > 50 IU/l
  3. For men: Throughout the duration of the treatment and for 3 months after the end of the protocol (i.e. one spermatogenesis cycle), sexual intercourse must always be protected by using a condom.

Exclusion Criteria:

* Pregnant or breast-feeding women or those of childbearing potential who are not using an effective method of contraception or the lack of protection during sexual intercourse in men.
* Patients who have already received treatment with thalidomide.
* Contraindication to thalidomide.
* Patient who has an absolute contraindication to dexamethasone.
* Patient with a history of deep vein thrombosis and who is not taking effective oral anticoagulation (the anticoagulant must be continued throughout the entire study).
* Performance index more than or equal to 3, unless the patient is bedridden as a result of the progress of the myeloma.
* Any situations that do not permit adequate follow-up of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2001-12-01 (Actual); Primary Completion 2005-10-01 (Actual); Study Completion 2006-04-01 (Actual)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
response rate | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim YAKOUB-AGHA, MD, Principal Investigator — CHRU LILLE
Locations (49):
- Belgium (2):
  - Hopital St Joseph, Gilly
  - UCL de Mont Godine, Yvoir
- France (47):
  - Chu D'Angers - Medecine D, Angers
  - Centre Hospitalier D'Annecy - Service d'oncohématologie, Annecy
  - Centre Hospitalier H. Duffaut - Hematologie, Avignon
  - HOPITAL JEAN MINJOZ - Médecine interne/Hématologie, Besançon
  - Centre Hospitalier de Blois - Unité d'Onco-Hématologie, Blois
  - Hopital Avicenne - Medecine Interne/Hematologie, Bobigny
  - Centre Hospitalier Du Dr Duschene - Hematologie, Boulogne-sur-Mer
  - Hopital Morvan - Service Hematologie, Brest
  - Polyclinique Du Parc - Hematologie, Caen
  - Centre François Baclesse, Caen
  - Centre Hospitalier - Service Hematologie, Chambéry
  - H.I.A. Percy Hematologie, Clamart
  - Centre Hospitalier General - Medecine Interne, Dunkirk
  - Hopital Albert Michallon - Hematologie, Grenoble
  - CENTRE HOSPITALIER DEPARTEMENTAL - Sce Médecine A, La Roche-sur-Yon
  - Centre Hospitalier La Rochelle - Unité d'Oncologie Médicale, La Rochelle
  - Centre Hospitalier - Service de Médecine 7, Laval
  - Clinique Victor Hugo, Le Mans
  - CHRU CLAUDE HURIEZ - Maladies du sang, Lille
  - Chu Edouard Herriot, Lyon
  - INSTITUT PAOLI CALMETTE - Unité transplantation, Marseille
  - CHR Hôp N.D. de Bon Secours - Service de Médecine A, Metz
  - Hopital Jacques Monod - Rhumatologie, Montivilliers
  - CHRU Hôtel Dieu, Service des Maladies du Sang, Nantes
  - Centre Lacassagne, Nice
  - Institut Curie - Service d'hématologie, Paris
  - HOPITAL ST ANTOINE - Maladies du Sang, Paris
  - Centre Hospitalier Général - Service d'Hématologie, Perpignan
  - Hopital Du Haut Leveque - Hematologie, Pessac
  - Centre Hospitalier de Lyon Sud, Pierre-Bénite
  - CHRU Jean Bernard - Hématologie, Poitiers
  - Centre Hospitalier Laennec - Service de Médecine A, Quimper
  - Hôpital Robert Debré - Hématologie, Reims
  - C.H.R. de Pontchaillou - Hématologie, Rennes
  - CHRU Hôpital Sud - Médecine Interne, Rennes
  - Centre Henri Becquerel - Service Hématologie, Rouen
  - C.H.U. de Saint Etienne - Hôpital Bellevue - Sce Rhumatologie, Saint-Etienne
  - Hôpital Nord - Hématologie, Saint-Etienne
  - CHU Hautepierre - Service Hématologie, Strasbourg
  - HOPITAL HAUTEPIERRE - Service Rhumatologie, Strasbourg
  - C.H.U. Rangueil - Service Rhumatologie, Toulouse
  - C.H.U. PURPAN - Service Hématologie, Toulouse
  - C.H.U. Bretonneau, Tours
  - Centre Hospitalier - Service de Rhumatologie, Tulle
  - Centre Hospitalier - Hématologie, Valence
  - CHU Hôpital Brabois - Médecine interne-Hématologie, Vandœuvre-lès-Nancy
  - Centre Hospitalier Chubert - Médecine Interne, Vannes

REFERENCES:
- [Background] Yakoub-Agha I, Mary JY, Hulin C, Doyen C, Marit G, Benboubker L, Voillat L, Moreau P, Berthou C, Stoppa AM, Maloisel F, Rodon P, Dib M, Pegourie B, Casassus P, Slama B, Damaj G, Zerbib R, Harousseau JL, Mohty M, Facon T; Intergroupe Francophone du Myelome (IFM). Low-dose vs. high-dose thalidomide for advanced multiple myeloma: a prospective trial from the Intergroupe Francophone du Myelome. Eur J Haematol. 2012 Mar;88(3):249-59. doi: 10.1111/j.1600-0609.2011.01729.x. Epub 2012 Jan 4. PMID 22023551